CLINICAL TRIAL: NCT05359029
Title: Duodenostomy on Foley and Gastroenteroanastomosis: Treatment of Second Duodenal Part Perforation.
Brief Title: Duodenostomy to Treat Duodenal Perforation
Status: Completed | Type: Observational
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Mario Pacilli, Principal Investigator, University of Foggia
Other Study IDs: UFoggia
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: The Focus of Study is to Elucidate Which Are the Factors Requiring the Duodenostomy and Which Postoperative Course is for These Patients
Keywords: Duodenostomy; duodenal perforation; emergency surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study the investigators focused on duodenal perforations, requiring a tube duodenostomy and have analyzed the main features, that have influenced the surgical choices. Five patients were enrolled. Most of duodenal perforations can successfully be managed by simple repair, while complicated procedures are needed for complex injuries. Tube duodenostomy is a damage control procedure, for large duodenal perforations when further repair techniques are not recommended due to the duodenal damage, hemodynamic instability of the patient or the absence of surgical expertise for complex reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* excessive size of perforation
* extreme presence of intra-abdominal infections.

Exclusion Criteria:

* patients treated by medical therapy, endoscopic techniques, o surgical approaches

Max Age: 89 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: In 2 cases a tube duodenostomy was executed, due to excessive size of perforation and extreme presence of intra-abdominal infections.
  In addition, other cases of duodenal injury due to other causes were treated, 3 of these requiring a tube duodenostomy approach.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Death of patient | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Di Foggia, Foggia, Italy

DOCUMENTS (1):
  • Study Protocol (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT05359029/Prot_001.pdf